CLINICAL TRIAL: NCT07406607
Title: The Effect of Presence of Father During Elective Cesarean Section Under Spinal Anesthesia on Parturient's Quality of Recovery
Brief Title: The Effect of Presence of Father in the Operating Room on Quality of Recovery of the Parturient
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Gamze Savci, Asst. Prof, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: E-11095095-050.04-253322
Record Dates: First submitted 2025-12-30; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Caesarean Section
Keywords: spinal anesthesia; obstetric quality of recovery; Caesarean section; surgeon comfort
MeSH Terms: interventions — Standard of Care; Operating Rooms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All the data collected will be assessed by a masked outcome assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partner Present (Experimental)
  Interventions: Other: Partner Presence in Operating Room
- Partner Absent (Active Comparator)
  Interventions: Other: Standard Care (No Partner Presence)

INTERVENTIONS:
Other: Standard Care (No Partner Presence) — The patient undergoes the elective cesarean section according to standard hospital protocols. The partner is not present in the operating room during the surgery.
  Arms: Partner Absent
Other: Partner Presence in Operating Room — The patient's partner is admitted to the operating room after sterile preparations are complete. The partner remains with the patient to provide physical and emotional support during the cesarean section operation
  Arms: Partner Present

SUMMARY:
The presence of a partner to support the mother during cesarean and vaginal deliveries is a well-established practice in most countries worldwide. It is evident that allowing the partner into the operating room during a cesarean section provides psychosocial benefits for both the mother and the partner. This study aims to investigate the effect of the presence of partner in the operating room on quality of recovery of parturients at the postoperative period.

DETAILED DESCRIPTION:
This prospective study evaluates the impact of the partner's presence in the operating room during elective cesarean sections on maternal anxiety, postoperative recovery, and surgeon stress levels. Patients are allocated into two groups: Partner Present and Partner Absent. Primary outcome is obstetric quality of recovery scale (ObsQoR 10) at the postoperative first day. Secondary outcomes include maternal pain (assessed via VAS at 6-hour intervals for the first 24 hours) and anxiety levels (STAI-T/S administered to couples preoperatively and STAI-S postoperatively) and ObsQoR-10 that will be evaluated at the postoperative 3rd and 7th days.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for an elective cesarean section.
* Patients and their partners must be literate in Turkish (able to read and write) to accurately complete the study questionnaires
* Patients and their partners must be willing and able to provide written informed consent
* Healthy pregnant women with no additional chronic or systemic diseases (comorbidities)
* The operating surgeon must have at least 5 years of professional experience and no chronic health conditions.

Exclusion Criteria:

* Patients undergoing emergency cesarean sections.
* Patients with any known chronic or systemic additional diseases
* Surgeons with any known chronic or systemic diseases.
* Individuals unable to read or understand the Turkish questionnaires (implied by the literacy requirement).
* Patients with American Society of Anesthesiologists (ASA) classification of 3 or more
* Patients with history of chronic pain, chronic use of analgesic drugs, or history of opioid or intravenous drug abuse
* Patients who have refused spinal anesthesia, or those in whom it is contraindicated.
* Pregnancy with preeclampsia or eclampsia
* Pregnancy with gestational diabetes mellitus or diabetes mellitus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-08 (Estimated)

PRIMARY OUTCOMES:
Obstetric Quality of Recovery-10 (ObsQoR-10) Score | Post-operative 24th hour,
  The ObsQoR-10 questionnaire will be used to assess the quality of maternal recovery after the cesarean section. The scale consists of 10 items, where patients rate each item from 0 (never) to 10 (always). Higher scores indicate a better quality of recovery.

SECONDARY OUTCOMES:
Surgeon's Physiological Stress Level (Heart Rate) | Intra-operative (during the entire duration of the cesarean section)
  The operating surgeon's heart rate variability will be recorded using a rhythm Holter device during the surgery. A heart rate exceeding 100 beats per minute (bpm) will be considered an indicator of increased stress.

OTHER OUTCOMES:
Maternal and Partner Anxiety Levels (STAI-T and STAI-S) | Pre-operative and Post-operative (within the first 6 hours)
  The State-Trait Anxiety Inventory (STAI) will be used to measure the patient's and partner's anxiety levels. Both the Trait (STAI-T) and State (STAI-S) components will be administered. Scores range from 20 to 80, with higher scores indicating greater anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)

REFERENCES:
- [Result] faruk